CLINICAL TRIAL: NCT01232595
Title: Multi-center, Randomized, Evaluator-blind, Active-controlled,Parallel-group Design to Determine Safety, Tolerability, and Efficacy of Multiple Daily Administration of LFF571 for 10 Days in Patients With Moderate Clostridium Difficile Infections
Brief Title: Safety and Efficacy of Multiple Daily Dosing of Oral LFF571 in Patients With Moderate Clostridium Difficile Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLFF571X2201; 2011-000947-26
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2015-03

CONDITIONS: Moderate Clostridium Difficile Infection
Keywords: Clostridium difficile,; C. difficile,; CDI,; Clostridium difficile-associated disease,; CDAD,; pseudomembranous colitis,; PMC,; antibiotic-associated diarrhea
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — LFF571; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- LFF571 (POC) (Experimental)
  Interventions: Drug: LFF571
- Vancomycin (POC) (Active Comparator)
  Interventions: Drug: Vancomycin (POC)
- LFF571 Dose level 1 (cohort 2) (Experimental)
  Interventions: Drug: LFF571
- LFF571 Dose level 2 (cohort 2) (Experimental)
  Interventions: Drug: LFF571
- LFF571 Dose level 3 (cohort 2) (Experimental)
  Interventions: Drug: LFF571
- LFF571 Dose level 4 (cohort 2) (Experimental)
  Interventions: Drug: LFF571

INTERVENTIONS:
Drug: LFF571
  Arms: LFF571 (POC); LFF571 Dose level 1 (cohort 2); LFF571 Dose level 2 (cohort 2); LFF571 Dose level 3 (cohort 2); LFF571 Dose level 4 (cohort 2)
Drug: Vancomycin (POC)
  Arms: Vancomycin (POC)

SUMMARY:
This study will assess the safety and efficacy of multiple daily dosing of oral LFF571 in patients who have moderate Clostridium difficile infections.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 90 years of age, inclusive.
* Diagnosed with primary episode or first relapse of moderate C. difficile infection.

Received ≤24 hours of therapy effective for C. difficile infection prior to enrollment.

Exclusion Criteria:

* Severe C. difficile infection
* Expected to require more than 10 days of C. difficile infection treatment.
* More than one prior episode of C. difficile infection within the prior 3 months.
* Use of anti-peristaltic drugs (including tincture of opium, metoclopramide, loperamide),, cholestyramine, or colestipol

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
POC: Difference in clinical response rate of LFF571 compared to vancomycin in patients with moderate C. difficile infections at day 12/13. | Day 12/13
POC: Safety and tolerability of LFF571 | Day 12/13
  Safety assessments will include vital signs, laboratory tests, electrocardiograms (ECG), pharmacokinetic (PK) samples and adverse events. (Cohorts 1 and 2)
POC:Clinical response rates (clinical cure) of patients with moderate C. difficile infections to different LFF571 dose regimens and total daily doses (cohort 2). | Day 12/13
  Clinical cure is resolution or improvement of symptoms and signs of C. difficile infection such that additional or alternative antimicrobial therapy or other theraperutic intervention is not needed. In addition, patient must have absence of fever for two consecutive days and <3 non-lliquid stools per day for two consecutive days
Cohort 2: Clinical response rate (clinical cure) of LFF571 in patients with mild and moderate C. difficile infections to different LFF571 dose regimens and total daily doses administered orally for 10 days | Day 12/13
  Clinical cure is resolution or improvement of symptoms and signs of C. difficile infection such that additional or alternative antimicrobial therapy or other theraperutic intervention is not needed. In addition, patient must have absence of fever for two consecutive days and <3 non-lliquid stools per day for two consecutive days.
Cohort 2: Dose-response relationship of different dose regimens and total daily dose s of LFF571 | Day 12/13
Cohort 2: Safety and tolerability of LFF571 dose regimens and total daily doses administered orally for 10 days to C. difficile infected patients. | Day 12/13
  Safety assessments will include vital signs, laboratory tests, electrocardiograms (ECG), pharmacokinetic (PK) samples and adverse events.

SECONDARY OUTCOMES:
POC: To evaluate the time to resolution of diarrhea during the treatment period for LFF571-treated patients (cohorts 1 and 2) | End of therapy
POC: To evaluate the relapse rate within 30 days following completion of LFF571-treated patients (cohort 1) | 30 days
POC: To evaluate the sustained response and relapse rate within 30 days following completion of different oral LFF571 dose regimens (cohort 2) | 30 days
POC: To evaluate the fecal concentrations of LFF571 following different LFF571 dose regimens (cohort 2) | 30 days
POC: To evaluate the serum concentrations of LFF571 following different LFF571 dose regimens. (cohort 2) | 30 days
Cohort 2: Time to resolution of diarrhea during the treatment period for oral LFF571 in C. difficile infected patients. | Day 12/13
Cohort 2: Serum concentrations of oral LFF571 following different dose regimens in C. difficile infected patients. | Day 12/13
Cohort 2: Fecal concentrations of LFF571 following different oral LFF571 dose regimens in C. Difficile infected patients. | Day 12/13
Cohort 2: Sustained response (sustained clinical cure) rate and clinical relapse rate at 30 days following completion of different oral LFF571 dose regimens. | 30 days
  Clinical cure is resolution or improvement of symptoms and signs of C. difficile infection such that additional or alternative antimicrobial therapy or other theraperutic intervention is not needed. In addition, patient must have absence of fever for two consecutive days and <3 non-lliquid stools per day for two consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (14):
  - Novartis Investigative Site, Palm Desert, California
  - Novartis Investigative Site, Bristol, Connecticut
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Idaho Falls, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Michigan City, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Butte, Montana
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, San Antonio, Texas
- Canada (4):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec

REFERENCES:
- [Derived] Mullane K, Lee C, Bressler A, Buitrago M, Weiss K, Dabovic K, Praestgaard J, Leeds JA, Blais J, Pertel P. Multicenter, randomized clinical trial to compare the safety and efficacy of LFF571 and vancomycin for Clostridium difficile infections. Antimicrob Agents Chemother. 2015 Mar;59(3):1435-40. doi: 10.1128/AAC.04251-14. Epub 2014 Dec 22. PMID 25534727
- [Derived] Bhansali SG, Mullane K, Ting LS, Leeds JA, Dabovic K, Praestgaard J, Pertel P. Pharmacokinetics of LFF571 and vancomycin in patients with moderate Clostridium difficile infections. Antimicrob Agents Chemother. 2015 Mar;59(3):1441-5. doi: 10.1128/AAC.04252-14. Epub 2014 Dec 22. PMID 25534724
- See also: Results for CLFF571X2201from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12263